CLINICAL TRIAL: NCT00344916
Title: NO-Synthesis in Patients With Liver Cirrhosis: Effect of L-NMMA on Renal Hemodynamics, Sodium Excretion and Plasma Levels of Vasoactive Hormones
Brief Title: Phase 1 Study of L-NMMA in Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MED.RES.HOS.1996.04.JNB
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2006-07-11 (Estimated); Status verified 2006-06

CONDITIONS: Liver Cirrhosis
Keywords: Renal hemodynamics; Nitric oxide
MeSH Terms: conditions — Liver Cirrhosis | interventions — omega-N-Methylarginine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Ng-monomethyl-L-arginine (drug)

SUMMARY:
Phase 1 study of the effects of nitric oxide inhibition with L-NMMA in patients with liver cirrhosis and healthy controls. It is hypothesized that nitric oxide availability is increased in liver cirrhosis.

DETAILED DESCRIPTION:
In a randomized, placebo controlled design the acute effects of Ng-monomethyl-L-arginine are studied on:

* renal hemodynamics (GFR and RPF)
* blood pressure and heart rate
* lithium clearance
* plasma levels of vasoactive hormones

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Age 20 to 60 years
* Both men and women
* Weight below 100 kg
* Normal clinical examination and laboratory screening
* Fertile women only if using contraception
* Informed consent according to the regulations of the local ethics committee

Liver cirrhosis

* Biopsy verified liver cirrhosis or clinical and laboratory signs of liver cirrhosis including hypoalbuminaemia, increased prothrombin time in combination with esophagusvarices or ascites
* P-creatinine < 250 µmol/L
* Age 20-60 years
* Both men and women
* Fertile women only if using contraception
* Body weight below 100 kg
* Informed consent according to the regulations of the local ethics committee

Exclusion Criteria:

Healthy controls

* History or clinical evidence of diseases of the heart and blood vessels, kidneys, liver and pancreas, endocrine organs, lungs, neoplastic disease, myocardial infarction or cerebrovascular insult as evaluated by clinical examination and laboratory screening
* Current medication
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances
* Donation of blood less than 1 month before the experiments

Liver cirrhosis

* Apart from liver cirrhosis no history of diseases of the heart and blood vessels, endocrine organs, lungs, myocardial infarction, cerebrovascular insult or neoplastic disease.
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark; Jesper N Bech, MD, Ph.d., Principal Investigator — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark